CLINICAL TRIAL: NCT06578286
Title: Evaluate the Efficacy and Safety of ARX788 in Patients With HER2-positive Advanced Breast Cancer Whose Disease Has Progressed Following T-DXd Therapy
Brief Title: ARX788 in HER2-positive Metastatic Breast Cancer Patients Who Were Previously Treated With T-DXd
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-Breast-10
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ARX788

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARX788 (Experimental): ARX788，1.5 mg/kg IV infusion on Day 1 of each 21-day treatment cycle
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — ARX788，1.5 mg/kg IV infusion on Day 1 of each 21-day treatment cycle

SUMMARY:
A single arm, phase 2 Study of ARX788 in HER2-positive metastatic breast cancer patients who were previously treated with T-DXd. The ARX788 will be administered every 3 weeks (Q3W) intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old (including upper and lower limits), male or female;
2. Unresectable locally advanced, recurrent or metastatic BC;
3. Tissue samples determined to be HER2 positive (defined as IHC3+ or FISH+);
4. Received T-DXd treatment in the advanced stage;
5. Adequate bone marrow, liver, kidney and coagulation function;
6. Voluntarily sign the informed consent, have good compliance and are willing to comply with the follow-up visit.

Exclusion Criteria:

1. With meningeal metastases or disseminated brain metastases or active brain metastases;
2. Has interstitial lung disease requiring steroid therapy, a history of drug-induced interstitial lung disease, a history of radiation pneumonitis, or any evidence indicating clinically active interstitial lung disease;
3. Has any eye disease that require medical intervention such as keratitis, corneal diseases or active eye infection;
4. Has cardiac insufficiency;
5. Has received any systemic anti-tumor therapy (with the exception of endocrine therapy, with an interval of at least 7 days) within 28 days (or at least 5 half-lives) before the first use of the investigational product;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | Until progression, assessed up to approximately 24 months
  The proportion of patients who have a CR or PR, as determined by the Investigator at local site per RECIST 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Baseline through end of study, assessed up to 24 months]
  The proportion of patients who have a CR or PR or SD, as determined by the Investigator at local site per RECIST 1.1.
Duration of relief (DOR) | Until progression, assessed up to approximately 24 months
  Time from the date of first documented response until the date of documented progression or death in the absence of disease progression
Progression-free survival (PFS) | Until progression or death, assessed up to approximately 36 months]
  Time to progression as assessed by the Investigator at local site per RECIST 1.1, or death due to any cause.
Overall survival (OS) | Until death, assessed up to approximately 50 months
  Time to death due to any cause
The number of subjects experiencing adverse event TEAEs | Up to follow-up period, approximately 50 months
  Occurrence of AEs according to CTCAE v5.0

IPD SHARING:
Plan to Share IPD: Undecided